CLINICAL TRIAL: NCT03606616
Title: A Prospective Feasibility Study Applying the ACOSOG Z0011 Criteria to Chinese Patients With Early Breast Cancer Undergoing Breast-conserving Surgery
Brief Title: Prospective Feasibility Study Applying the ACOSOG Z0011 Criteria to Chinese Patients
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Peng Yuan, Peking University People's Hospital Breast Center, Peking University People's Hospital
Other Study IDs: ACOSOGZ0011CH
Record Dates: First submitted 2018-07-20; First posted 2018-07-31 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer; Sentinel Lymph Node; Local Recurrence of Malignant Tumor of Breast
Keywords: ACOSOG Z0011; Chinese breast cancer; sentinel lymph node; overall survival; disease-free survival
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACOSOG Z0011 no further ALND arm: patients meeting the criteria for ACOSOG Z0011 trial inclusion：histologically confirmed invasive breast cancer;clinical T1/T2;breast conserving surgery；1 or 2 positive sentinel lymph nodes; Whole-breast RT planned; no preoperative chemotherapy
  Interventions: Procedure: no further ALND arm

INTERVENTIONS:
Procedure: no further ALND arm — Patients meeting the Z0011 inclusion criteria to receive no additional ALND

SUMMARY:
In patients undergoing breast-conserving surgery and having positive sentinel lymph nodes (SLNs), the ACOSOG Z0011 trial showed equivalent overall survival(OS) and disease-free survival(DFS) outcomes for patients receiving SLN dissection (SLND) alone and those receiving axillary lymph node dissection (ALND). We conducted a prospective single-arm study to confirm the applicability of the Z0011 criteria to Chinese patients with breast cancer.

DETAILED DESCRIPTION:
The American College of Surgeons Oncology Group (ACOSOG) Z0011 trial demonstrated that in clinically node-negative women with T1 or T2 invasive breast cancer, who underwent breast-conserving surgery (BCT) with whole breast irradiation (WBRT), had excellent local control and survival with SLND alone, even if metastases were found in 1 or 2 SLNs. Recently, the long-term follow-up data of the Z0011 study were reported, which demonstrated that the 10-year OS for patients receiving SLND alone was not inferior to that for those receiving ALND.

This breakthrough result of the Z0011 study led to a change in clinical practice regarding the standard management of axillary lymph nodes in patients with breast cancer.

However, these validation data have been generated in Western populations. As the socio-economic profile, life style and culture of Asian are substantially different from those of Western, and genetic backgrounds vary to some extent, it remains unclear whether results similar to those of the Z0011 study could be achieved in a Chinese breast cancer population. In the present study, we prospectively applied the Z0011 eligibility criteria to Chinese patients with clinically node-negative breast cancer undergoing BCT, with planned RT. The purpose of this study is the clinicopathological relevance of the Z0011 findings for Chinese patients with breast cancer, and to verify the feasibility of using the Z0011 criteria to avoid ALND after positive SLN findings.

This is a prospective single-arm study, enrolled patients meeting Z0011 inclusion criteria and providing consent to receive no additional ALND. Overall survival is the primary end point, disease-free survival and occurrence of surgical morbidities a secondary end point.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed invasive breast cancer T1 or T2 tumor 1 or 2 positive sentinel lymph nodes breast-conserving surgery whole-breast RT planned

Exclusion Criteria:

* preoperative therapy 3 or more positive sentinel lymph nodes patients undergoing additional mastectomy due to positive surgical margins

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: histologically confirmed invasive breast cancer patients, who meeting the critiera of Z0011 inclusion: T1 or T2 tumor,1 or 2 positive sentinel lymph nodes,breast-conserving surgery and whole-breast RT planned is enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
overall survival | 5 years
  the time from surgery until death from any cause

SECONDARY OUTCOMES:
disease-free survival | 5 years
  the time from surgery to death or first documented recurrence of breast cancer
occurrence of surgical morbidities | 5 years
  edema，limited activity or pain on surgical side upper limb

CONTACTS AND LOCATIONS:
Overall Officials: shu wang, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking university people's hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Peng Y, Liu M, Li X, Tong F, Cao Y, Liu P, Zhou B, Liu H, Cheng L, Guo J, Xie F, Yang H, Wang S, Wang C, Chen Y, Wang S. Application of the ACOSOG Z0011 criteria to Chinese patients with breast cancer: a prospective study. World J Surg Oncol. 2021 Apr 20;19(1):128. doi: 10.1186/s12957-021-02242-1. PMID 33879180